CLINICAL TRIAL: NCT00619047
Title: The Role of Impact Activity in Peripubertal Bone Accrual
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Tamara A. Scerpella, MD, SUNY Upstate Medical University
Other Study IDs: Bone Density Study
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Bone Mineral Density

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation

SUMMARY:
Osteoporosis has been established as a major public health problem, primarily effecting women. The attainment of maximal peak bone mass is crucial in the prevention of osteoporosis, yet little is known about the specifics of bone accrual. Physical activity has been identified as an important modifiable factor controlling bone accrual. It is has been shown that increased activity during peri-pubertal years increase bone mineral content during adulthood. Thus, strategies designed to increase peak bone mass should target the peri-pubertal years of critical bone acquisition.

Hypothesis 1a: The amount of bone mineral accrued during the peri-pubertal years is greater in girls who engage in impact activity than in those who do not.

Hypothesis 1b: The positive effects of impact activity on bone accrual are maintained after cessation of the activity, resulting in greater bone mineral density in girls who participate in impact activity during a portion of the peri-pubertal years than in those who never participated in impact activity.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 10-12 will be asked to participate

Ages: 10 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects were recruited into the following three groups based on their exposure to gymnastic activity. A) control, no gymnastic activity. B)retired gymnasts, who participated at study onset, but stopped gymnastics activity during the course of the study. C) active gymnast, who continues participation in gymnastics throughout the duration of the study.
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2002-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara A Scerpella, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- Institute for Human Performance, Syracuse, New York, United States